CLINICAL TRIAL: NCT04383418
Title: Study on Efficacy and Safety of Dexmedetomidine Hydrochloride Nasal Spray for Preoperative Sedation in Adults
Brief Title: A Trial of Dexmedetomidine Hydrochloride Nasal Spray in Preoperative Sedation of Adults
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR0171401-301
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Preoperative Sedation

STUDY DESIGN:
Intervention Model Description: Dexmedetomidine hydrochloride nasal spray compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose group (Experimental): In the low dose group, 36 subjects will receive a low dose of dexmedetomidine nasal spray.
  Interventions: Drug: dexmedetomidine nasal spray
- Low dose group (Experimental): In the high dose group, 36 subjects will receive a high dose of dexmedetomidine nasal spray.
  Interventions: Drug: dexmedetomidine nasal spray
- Placebo group (Placebo Comparator): In the placebo group，36 subjects will receive dexmedetomidine hydrochloride nasal spray blank preparation.
  Interventions: Drug: dexmedetomidine hydrochloride nasal spray blank preparation

INTERVENTIONS:
Drug: dexmedetomidine nasal spray — dexmedetomidine nasal spray
  Arms: High dose group; Low dose group
Drug: dexmedetomidine hydrochloride nasal spray blank preparation — dexmedetomidine hydrochloride nasal spray blank preparation
  Arms: Placebo group

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of dexmedetomidine hydrochloride nasal spray for preoperative sedation in adults. To explore the reasonable dosage of dexmedetomidine hydrochloride nasal spray for preoperative sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective general anesthesia surgery
3. Male or female
4. Meet the weight standard
5. Conform to the ASA Physical Status Classification

Exclusion Criteria:

1. Not suitable for nasal spray
2. Subjects who had received general anesthesia
3. Subjects with a history of myocardial infarction or unstable angina pectoris
4. Subjects with atrioventricular block or cardiac insufficiency
5. Subjects with a history of ischemic stroke or transient ischemic attack
6. Subjects with poor blood pressure control after medication
7. Subjects with abnormal clotting function
8. Subjects with a history of mental illness and a history of cognitive impairment epilepsy
9. Subjects with a history or possibility of a difficult airway
10. Subject with a history of substance abuse and drug abuse
11. Adrenoceptor agonists or antagonists were used before randomization
12. Abnormal values in the laboratory
13. Thyroid dysfunction
14. Allergic to a drug ingredient or component
15. Pregnant or nursing women
16. No birth control during the specified period of time
17. Participated in clinical trials of other drugs (received experimental drugs)
18. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-05-31 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-09-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who meet the Ramsay sedation score of 3 at least once within 45 minutes | 0 minute to 45 minutes after administration
  Evaluated with Ramsay sedation scale Score Response
  1. Anxious or restless or both
  2. Cooperative, orientated and tranquil
  3. Responding to commands
  4. Brisk response to stimulus
  5. Sluggish response to stimulus
  6. No response to stimulus

SECONDARY OUTCOMES:
Total consumption of propofol during bispectral index reaches 60 for the first time | The bispectral index reaches 60 for the first time during intraoperative
  Total consumption of propofol during bispectral index reaches 60 for the first time
Total consumption of propofol during general anesthesia | From the beginning of anesthesia to the end of surgical operation up to 4 hours
  Total consumption of propofol during general anesthesia
Total consumption of opioid analgesic during bispectral index reaches 60 for the first time | The bispectral index reaches 60 for the first time during intraoperative
  Total consumption of opioid analgesic during bispectral index reaches 60 for the first time
Total consumption of opioid analgesic during general anesthesia | From the beginning of anesthesia to the end of surgical operation up to 4 hours
  Total consumption of opioid analgesic during general anesthesia
The BIS value for the Ramsay sedation score of 3 for the first time after administration | The Ramsay sedation score of 3 for the first time during intraoperative
  The BIS value for the Ramsay sedation score of 3 for the first time after administration
Anesthesiologist satisfaction rating | At the end of surgery when the patient recovers from anesthesia
  The anesthesiologist satisfaction rating is a scale of 0 to 10, satisfaction defined as a scale of 10, dissatisfaction defined as a scale of 0.
Subjects' satisfaction rating | From the end of surgical operation up to 24 hours
  The subjects' satisfaction rating is a scale of 0 to 10, satisfaction defined as a scale of 10, dissatisfaction defined as a scale of 0.

CONTACTS AND LOCATIONS:
Overall Officials: Changhong Miao, PhD, Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China